CLINICAL TRIAL: NCT06327581
Title: Comparative Study of Combined Microneedling With Either 1% Lactic Acid Solution or Vitamin D3 or Triamcinolone Acetonide in The Treatment of Alopecia Areata
Brief Title: Combined Microneedling With Either 1% Lactic Acid Solution or Vitamin D3 or Triamcinolone Acetonide in The Treatment of Alopecia Areata
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Rana Ehab, lecturer of dermatology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101005
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Lactic Acid; Triamcinolone Acetonide; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- lactic acid group (Experimental): · First group (A): 22 AA patients will be treated with MN combined with lactic acid solution 1%.
  Interventions: Drug: Lactic Acid
- vitamin d3 (Experimental): · Second group (B):22 AA patients will be treated with MN combined with topical application of vitamin D3 (an aqueous preparation of cholecalciferol (Devarol® ampoule 200 000 IU/2 ml, Memphis, Egypt) (2.5 mg/ ml), The maximum total amount of vitamin D3 injected into a patient in every session will be 2.5 mg (1 ml)
  Interventions: Drug: vit D
- triamcinolone acetonide group (Experimental): · Third group (C): 22 AA patients will be treated with MN combined with triamcinolone acetonide injectable suspension (Epirelefan®, 40mg/ ml, Eipico, Egypt) (10 mg/ml) will be used in a dose of 0.1 ml/cm2 area
  Interventions: Drug: Triamcinolone Acetonide
- saline (Experimental): · Fourth group (D): 22 AA patients will be treated with MN combined with normal saline 0.9%
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lactic Acid — patients will be treated with MN combined with lactic acid solution 1%.
  Arms: lactic acid group
Drug: vit D — patients will be treated with MN combined with topical application of vitamin D3 (an aqueous preparation of cholecalciferol (2.5 mg/ ml), The maximum total amount of vitamin D3 injected into a patient in every session will be 2.5 mg (1 ml)
  Arms: vitamin d3
Drug: Triamcinolone Acetonide — patients will be treated with MN combined with triamcinolone acetonide injectable suspension (Epirelefan®, 40mg/ ml, Eipico, Egypt) (10 mg/ml) will be used in a dose of 0.1 ml/cm2 area
  Arms: triamcinolone acetonide group
Drug: Saline — patients will be treated with MN combined with normal saline 0.9%
  Arms: saline

SUMMARY:
Alopecia areata (AA) is an immunologically mediated disease characterized by non-scarring hair loss (Madni and Shapiro, 2000). AA is presented by rapid and complete hair loss in one or more round or oval patches, usually on the scalp, beard area, eyebrows, eyelashes, and less commonly, on other hairy areas of the body (Berker et al., 2010 and James et al., 2011) Alopecia areata is a T-cell-mediated autoimmune disease. There is a complicated interplay between loss of immune privilege in the hair follicle, autoimmune-mediated hair follicle damage, and activation of inflammatory pathways that have been argued to explain the development of this disorder, but the exact pathophysiology of AA remains unknown. Hair follicles are infiltrated by autoreactive CD8 and CD4 T lymphocytes, which attack hair follicle-derived autoantigens while sparing the stem compartment (Rajabi et al., 2018).

Alopecia areata can be treated with topical and/or intralesional corticosteroids, which are the treatment of choice. Anthralin, minoxidil, coal tar, and topical immunotherapy are examples of other topical treatments. Systemic immunosuppressants such as cyclosporine, systemic steroids, Janus kinase inhibitors, and methotrexate may be considered in severe resistant cases (lee and lee, 2017).

Intralesional triamcinolone acetonide is preferred in cases of AA , as it is well known as anti-inflammatory and interferes with local immunity of the skin, which helps in the recovery of the disease, but if used in wrong technique or given in a high dose, it might cause all the side effects of corticosteroid, especially skin atrophy (Berker et al., 2010).

Lactic acid is a member of alpha-hydroxy acids. It has been used in the treatment of many skin diseases, like AA and vitiligo. Lactic acid stimulates spontaneous secretion of vascular endothelial growth factor (VEGF) by human reconstructed epidermis. VEGF is an angiogenic cytokine involved in angiogenesis and wound healing and stimulates the growth of hair follicles resulting in recovery of AA. Other studies suggest that lactic acid may act through its irritant effect (Al-Tammimy, 2005).

Vitamin D interacts with the innate and adaptive immune systems in a variety of ways, the majority of which contribute to its downregulation (Nancy and Yehuda, 2009). It has a powerful effect on T and B lymphocytes, influencing their activation responses (Arnson et al., 2007).

All cells of the immune system express 1,25-dihydroxyvitamin D3 receptors (VDRs) and are therefore vulnerable to calcitriol-mediated modulation. Vitamin D3 has the ability to influence the migration and maturation of different dendritic cell subtypes and their production of chemokines and cytokines, giving them an immunoregulatory and tolerogenic role (Illescas-Montes et al., 2019) It has been shown that VDRs are highly expressed in the keratinocytes of human hair follicles and the absence of their expression is associated with reduced hair follicle growth and epidermal differentiation. Reduced VDR expression in the hair follicles of affected areas has also been observed in studies of AA patients' scalp (Çerman et al., 2015).

Microneedling (MN) is a technique that comprises puncturing the skin repeatedly with sterile microneedles (Iriarte et al., 2017). It promotes hair regeneration by triggering stem cells in the hair bulge, which results in the generation of growth factors. It also improves blood circulation to the hair follicles and influences the local immune cells (Chandrashekar et al., 2014). Moreover, combining MN with applied topical drugs facilitates their absorption through the microchannels created within the epidermis (Fertig et al., 2018).

DETAILED DESCRIPTION:
Patients in all groups will be subjected to microneedling (MN) using a dermapen "Dr.Pen") with adjustable needle length ranging from 1.5 to 2 mm, using the highest speed level (4-5). First, topical anesthetic cream will be applied. Then, they will be stroked by dermapen diagonally, vertically, and horizontally in a repeated manner until pinpoint bleeding appears which will be regarded as an endpoint.

* First group (A): 22 AA patients will be treated with MN combined with lactic acid solution 1%. (Sharquis et al., 2015).
* Second group (B): 22 AA patients will be treated with MN combined with topical application of vitamin D3 (an aqueous preparation of cholecalciferol (Devarol® ampoule 200 000 IU/2 ml, Memphis, Egypt) (2.5 mg/ ml), The maximum total amount of vitamin D3 injected into a patient in every session will be 2.5 mg (1 ml) (Ali et al., 2023).
* Third group (C): 22 AA patients will be treated with MN combined with triamcinolone acetonide injectable suspension (Epirelefan®, 40mg/ ml, Eipico, Egypt) (10 mg/ml) will be used in a dose of 0.1 ml/cm2 area (Arora et al., 2022).
* Fourth group (D): 22 AA patients will be treated with MN combined with normal saline 0.9% In all groups, sessions were done every 2 weeks for a maximum of six sessions. V. Photographs will be taken by (Iphone 13 pro max Camera) before, during and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* · Age ≥ 16 years old with localized patchy AA (up to 6 cm in diameter).

  * Patients of both sexes
  * Willing to participate in the study and to sign an informed consent.

Exclusion Criteria:

* · Patients who received systemic or topical treatment for AA in the last 3 months prior to the start of the study

  * Patients with Alopecia totalis, universalis, ophiasis, or sisaipho
  * Pregnant or lactating females
  * Patients who had bleeding or coagulation disorders
  * Immunocompromised patients
  * Patients with known history of hypersensitivity to vit D
  * Patients taking vitamin D supplements in the last 6 months.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — more than 16 years old
Enrollment: 88 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
hair regrowth improvement assessed by SALT score and percaentage of hair growth | 3 months
  Clinical scoring: The evaluation of therapeutic response will be carried out by three blinded investigators to determine the percentage of improvement as follows using SALT score and percentage of hair growth (A0 = no change or further hair loss, A1=1-24% regrowth, A2= 25-49%, A3=50-74%, A4= 75-99%, A5= 100% regrowth

CONTACTS AND LOCATIONS:
Overall Officials: rana ehab, md, Principal Investigator — Zagazig University
Locations (1):
- Rana Ehab, Zagazig, Egypt